CLINICAL TRIAL: NCT01573520
Title: A Randomized Trial Comparing an Integrated Care Approach Using Electronic Cinacalcet Adherence Data Versus Usual Care to Improve Secondary Hyperparathyroidism in Hemodialysis Patients
Brief Title: Treatment Adhesion in Dialysis Patients Treated With Cinacalcet
Acronym: MEMS-cinac
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michel Burnier (Other)
Responsible Party: Sponsor-Investigator, Michel Burnier, Centre Hospitalier Universitaire Vaudois, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 268/09
Record Dates: First submitted 2012-03-23; First posted 2012-04-09 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Hyperparathyroidism; Chronic Kidney Disease
Keywords: compliance; dialysis; hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism; Renal Insufficiency, Chronic; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention)
- adherence intervention arm (Active Comparator): Monitoring drug adherence to guide treatment
  Interventions: Other: Monitoring of drug adherence

INTERVENTIONS:
Other: Monitoring of drug adherence — In the IC group, biological and drug adherence results are shown and discussed through a nephrologists leaded semi-structured motivation interviews at interval of 2 months.
  Other Names: Compliance monitoring
  Arms: adherence intervention arm

SUMMARY:
Controlling secondary hyperparathyroidism (sHPT) in maintenance hemodialysis (MHD) patients is cumbersome, partly due to patient's non-adherence to prescribed drugs.

The main objective of this study was to assess whether an integrated care (IC) approach, in which adherence data are integrated in the decisional process, led to improved therapeutic control of secondary hyperparathyroidsm and higher percentages of bone metabolism targets as compared to a usual care (UC) approach, in which biological values represent the main stem of the decisional process.

The predefined hypothesis was that patients of the IC group should reach the iPTH targets using 25% less doses of cinacalcet at 6 months than those of the UC group.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients on hemodialysis since more than 3 months
* Patients with secondary hyperparathyroidism treated with Cinacalcet-HCl at a stable dose (30mg/day or more) for at least 1 month before enrolment and indication to Cinacalcet-HCL therapy (iPTH in target values or over target values)
* Patients with secondary hyperparathyroidism with indication to be treated with Cinacalcet-HCL (iPTH ≥ locally pre-defined targets). In this case, patients should be treated at least 1 month with stable dose Cinacalcet-HCL before enrolment

Exclusion Criteria:

* Intolerance to Cincalcet-HCL
* Inability to understand the protocol
* Mental diseases
* Patients suffering from cancer or having a short life expectancy (<6 months)
* Patients planned for a parathyroidectomy
* Patients having had a parathyroidectomy
* Patient already enrolled in a Cinacalcet-HCL protocol
* Symptomatic hypocalcaemia or total serum calcium < 1.87 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in cinacalcet dose at 6 months | baseline and 6 months
  * (6-months dose - baseline dose)/ baseline dose %
  * dose expressed in mg/d

SECONDARY OUTCOMES:
absolute change from baseline in iPTH at 6 months | baseline and 6 months
  * 6-months iPTH - baseline iPTH
  * iPTH (=intact parathyroid hormone), unit ng/l

CONTACTS AND LOCATIONS:
Overall Officials: Michel Burnier, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland